CLINICAL TRIAL: NCT05231889
Title: Radifocus (Terumo) Versus Silverway (Asahi) to Deliver Catheters During Cardiac Catheterization
Acronym: RADVES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Principal Investigator, Koen Ameloot, Medical doctor, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Z-2021119
Record Dates: First submitted 2022-01-29; First posted 2022-02-09 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Anomalies Vascular
Keywords: Cardiac catheterization; Radifocus guide wire; Silverway guide wire
MeSH Terms: conditions — Vascular Malformations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Below the shoulder vascular anomaly (Placebo Comparator): If the standard J-tip guidewire does not cross a vascular anomaly located below the shoulder
  Interventions: Device: Radifocus guidewire
- Above the shoulder vascular anomaly (Active Comparator): If the standard J-tip guidewire does not cross a vascular anomaly located above the shoulder
  Interventions: Device: Silverway guidewire

INTERVENTIONS:
Device: Silverway guidewire — The Silverway guidewire is a newly developed guidewire to overcome the problems the Radifocus guidewire has
  Arms: Above the shoulder vascular anomaly
Device: Radifocus guidewire — The Radifocus guidewire is a hydrophilic coated guidewire that is used when a standard J-tip guidewire does not cross a vascular anomaly
  Arms: Below the shoulder vascular anomaly

SUMMARY:
In some cases the standard J-tip guidewire cannot deliver the catheter into the aortic root, because of arterial loops or spasm. In these cases a hydrophilic guidewire (Terumo) gives the right lubricity and good shape retention to guide the catheter through the artery. However, the Terumo wire does not give much torque and could therefore easily penetrate side branches and cause dissection or perforation. The latest Silverway guidewire has some new advantages which is easier to guide and could cause less complications while faster delivery of catheters to the aortic valve. The investigators aim to compare both guide wires.

DETAILED DESCRIPTION:
During cardiac catheterization a catheter is threaded through the radial arteries to the aortic root with the support of a guide wire. The standard workhorse to deliver the catheter is a J-tip guidewire (spring coil wire). However, in patients with arterial tortuosity or spasm, this guidewire has low lubricity and no torque to direct the catheter because the outer coil and core are not connected together.

If this problem is encountered, interventional cardiologists will use a hydrophilic polymer-coated guide wire. Up to date there are several hydrophilic coated guide wires available. One of these is the Radifocus Guide Wire M (Terumo, Japan). Although it has better torque transmission than the spring wire, it still has low torque transmission due to a Nitinol core structure, is less supportive and can easily enter side branches because of the high lubricity and therefore might cause dissections or perforations.

In some cases, coronary angioplasty guide wires are needed to negotiate a highly tortuous artery, but they lack the support to advance the catheter.

Recently, the Silverway Guide Wire has been created (Asahi Intecc Co, LTD., Japan) to overcome the problems that a spring- and polymer wire have. Features that this new guide wire provide is hybrid coating and ACT ONE technology that connects the wire core and coil to ensure one to one torque transmission The investigators aim to compare both guide wires in deliverability, workability and complication rate.

ELIGIBILITY:
Inclusion Criteria:

* Indication for radial artery access for diagnostic cardiac catheterization
* Being able to receive the per standard protocol Verapamil and Nitroglycerin administration via radial artery
* Not able to deliver a diagnostic or guiding catheter to the aortic root by means of the standard J tip wire
* No signs of early complication after initial attempt with the J tip wire such as dissection, perforation or hematoma
* Age ≥ 18 years

Exclusion Criteria:

* Femoral or brachial artery access
* Patients with known CREST syndrome or other forms of scleroderma
* Emergent indication for cardiac catheterization such as an acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-07-12 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
Time in seconds from introduction to aortic root | During procedure
  Measuring time from entering the guidewire in the catheter to delivery of the catheter to the aortic root (in seconds)

SECONDARY OUTCOMES:
The ability of the study wire to deliver the catheter to the aortic root | During procedure
  If the study wire is able to deliver the catheter to the aortic root
Change of access site | During procedure
  Is change of access site necessary?
Interventional cardiologists' survey of grading parameters working with the guide wire | Directly after procedure. Scale: not satisfactory (1) - somewhat satisfactory (2) - satisfactory (3)
  The interventional cardiologist who used the study wire must fill up a survey after procedure to grade the workability and deliverability of the study wire

CONTACTS AND LOCATIONS:
Overall Officials: Koen Ameloot, Dr., Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No